CLINICAL TRIAL: NCT05574504
Title: Phase II Trial of Lurbinectedin Combined With Avelumab as Switch Maintenance Firstline Therapy for Metastatic Urothelial Carcinoma With Stable or Responding Disease Following Platinum-based Chemotherapy
Brief Title: Phase II Trial of Lurbinectedin Combined With Avelumab as Switch Maintenance Firstline Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Decision based on no enrollment
Sponsor: AdventHealth (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Guru Sonpavde, Study Principal Investigator, AdventHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VT# IST-21-11721
Record Dates: First submitted 2022-09-19; First posted 2022-10-10 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Cancer; Urothelial Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Transitional Cell | interventions — avelumab; PM 01183

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- avelumab (PD-L1 inhibitor immunotherapy) + lurbinectedin (Experimental): Phase II trial is designed to evaluate the combination of avelumab (800 mg IV every 2 weeks-(days 1,15, and 29 every 6 week cycle ) and lurbinectedin (3·2 mg/m2 lurbinectedin administered as a 1-h intravenous infusion once every 3 weeks-day 1 and 22 every 6 week cycle ) for those with stable or responding disease following 4-6 cycles of platinum-based firstline chemotherapy for mUC with stable or responding disease following 4-6 cycles of platinum-based firstline chemotherapy for mUC.
  Interventions: Drug: avelumab (PD-L1 inhibitor immunotherapy) + lurbinectedin

INTERVENTIONS:
Drug: avelumab (PD-L1 inhibitor immunotherapy) + lurbinectedin — Avelumab 800 mg IV q 2 weeks (days 1,15, and 29 every 6 week cycle ) (premedication includes a H1 blocker, H2 blocker and Tylenol) Lurbinectedin 3.2 mg/m2 administered as a 1-h intravenous infusion once every 3 weeks (day 1 and 22 every 6 week cycle )
  1 cycle= 6 weeks
  Premedication for lurbinectedin:
  * Corticosteroids (dexamethasone 8 mg intravenously or equivalent)
  * Serotonin antagonists (ondansetron 8 mg intravenously or equivalent) Granulocyte-colony stimulating factor (G-CSF) or equivalent per ASCO guidelines per investigator discretion

SUMMARY:
A nonrandomized phase II trial is proposed combining avelumab (PD-L1 inhibitor immunotherapy) + lurbinectedin as switch maintenance therapy for mUC following stable or responding disease on 4-6 cycles of first line platinum-based chemotherapy

DETAILED DESCRIPTION:
The purpose of this research is to study benefit of the combination of lurbinectedin chemotherapy with maintenance avelumab immunotherapy in patients with advanced cancer of the urinary tract who have completed platinum-based chemotherapy. Avelumab alone is the usual approach and is already approved by the US FDA for the treatments of patients with this type of cancer. Lurbinectedin is approved for a type of lung cancer, but is not approved for urinary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligibility should be reviewed and documented by an appropriate member of the investigator's study team before patients are included in the study. Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

  1. Diagnosis:

     1. Histologically confirmed, unresectable locally advanced or metastatic predominant transitional cell carcinoma of the urothelium.
     2. Documented Stage IV disease (T4b, N0, M0; any T, N1-N3, M0; any T, any N, M1) at the start of first-line chemotherapy.
     3. Measurable disease prior to the start of first-line chemotherapy by RECIST v1.1.
  2. Prior first-line chemotherapy must have completed 4-10 weeks before registration and consisted of at least 4 cycles and no more than 6 cycles of platinum-based chemotherapy. No other chemotherapy regimens are allowed in this study 3. Patients without progressive disease as per RECIST v1.1 guidelines (ie, with an ongoing CR, PR, or SD) following completion of 4 to 6 cycles of first-line chemotherapy.

     1. Eligibility based on this criterion will be determined by investigator review of pre-chemotherapy and post-chemotherapy radiological assessments (CT/MRI scans)

  4. Tumor samples: Provision of a recent formalin-fixed, paraffin-embedded (FFPE) tumor tissue block or slides from the most recent primary or metastatic tumor biopsy or resection obtained prior to treatment with first line chemotherapy is desirable (but not mandatory). If an FFPE tissue block cannot be provided, 15 unstained slides of 5 µM sections (10 minimum) will be acceptable.

  5. Evidence of a signed and dated informed consent document indicating that the patient (or a legally acceptable representative, as allowed by local guideline/practice) has been informed of all pertinent aspects of the study. 6. Patients who are willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

  7. Age >18 years. 8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2. 9. Adequate bone marrow function, including:
  1. Absolute neutrophil count (ANC) ≥1,500/mm3 or ≥1.5 x 109/L;
  2. Platelets ≥100,000/mm3 or ≥100 x 109/L;
  3. Hemoglobin ≥8 g/dL (may have been transfused). 10. Adequate renal function, defined as estimated creatinine clearance ≥30 mL/min as calculated using the Cockcroft-Gault equation.

     11. Adequate liver function, including: a. Total serum bilirubin ≥1.5 x upper limit of normal (ULN); b. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥2.5 x ULN.

     12. Serum pregnancy test (for females of childbearing potential) negative at screening.

     13. Male patients able to father children and female patients of childbearing potential and at risk for pregnancy must agree to use 2 highly effective methods of contraception throughout the study and for at least 60 days after the last dose of assigned treatment

     Exclusion Criteria:
* Patients with any of the following characteristics/conditions will not be included in the study:

  1. Patients whose disease progressed by RECIST v1.1 on or after first-line chemotherapy for urothelial cancer.
  2. Prior adjuvant or neoadjuvant therapy within 12 months of registration
  3. Prior immunotherapy with IL-2, PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or CTLA-4 antibody (including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
  4. Major surgery <4 weeks or major radiation therapy <2 weeks prior to randomization. Prior palliative radiotherapy (10 fractions) to metastatic lesion(s) is permitted, provided it has been completed at least 48 hours prior to patient randomization.
  5. Patients with known symptomatic central nervous system (CNS) metastases requiring steroids. Patients with previously diagnosed CNS metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to randomization, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable.
  6. Persisting toxicity related to prior therapy NCI CTCAE v5.0 Grade >1; however, sensory neuropathy Grade ≤2 is acceptable.
  7. Diagnosis of any other malignancy within 2 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix, or low-grade (Gleason ≤6) prostate cancer on surveillance without any plans for treatment intervention (eg, surgery, radiation, or castration), or any other cancer that is felt by the PI to be clinically insignificant not requiring systemic therapy in future.
  8. Participation in other studies involving investigational drug(s) within 4 weeks prior to randomization. Observational studies are permitted.
  9. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
  10. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, deep vein thrombosis, or symptomatic pulmonary embolism.
  11. Active infection requiring systemic therapy.
  12. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥3), any history of anaphylaxis, or uncontrolled asthma (ie, 3 or more features of asthma symptom control per the Global Initiative for Asthma 2015).
  13. Known prior or suspected hypersensitivity to study drugs or any component in their formulations.
  14. Current or prior use of immunosuppressive medication within 7 days prior to registration, EXCEPT the following:

      1. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection);
      2. Systemic corticosteroids at physiologic doses equivalent;
      3. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
  15. Diagnosis of prior immunodeficiency or organ transplant requiring immunosuppressive therapy, or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
  16. Any test for hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating acute or chronic infection.
  17. Vaccination within 4 weeks of the first dose of study treatment and while on trial is prohibited except for administration of inactivate vaccines (for example, inactivated influenza vaccines).
  18. Patients who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or patients who are Jazz Pharma employees directly involved in the conduct of the study.
  19. Pregnant female patients; breastfeeding female patients; male patients able to father children, and female patients of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in the protocol for the duration of the study and for at least 60 days after the last dose of investigational product.
  20. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, and pneumonitis; psychiatric condition including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
The combination of lurbinectedin chemotherapy with maintenance avelumab immunotherapy in patients with advanced cancer of the urinary tract | 32 months
  The primary objective of this study is to evaluate the progression-free survival (PFS) with switch maintenance combination of avelumab and lurbinectedin in patients with metastatic urothelial carcinoma with stable or responding disease with 4-6 cycles of platinum-based chemotherapy.

SECONDARY OUTCOMES:
The secondary objectives of this study are to assess: | 32 months
  A. Objective response rate (ORR) for those with measurable disease. B. Duration of response (DOR)
  Response will be measured using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
  Duration of Response is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented, or death due to any cause
Overall Survival (OS) | 32 months
  Overall Survival (OS) is defined as the time from treatment initiation to death due to any cause or censored at date last known alive.
Toxicities, associated with the combination treatment | 32 months
  For safety and tolerability, all adverse events will be graded and analyzed using CTCAE version 5.0. The worst grade will be used if any toxicity event is reported multiple times on the same participant. Any adverse events resulting in discontinuation, dose modification, and/or dosing interruption, and/or treatment delay of drug will also be summarized.

CONTACTS AND LOCATIONS:
Locations (1):
- AdventHealth Cancer Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No